CLINICAL TRIAL: NCT00026247
Title: A Phase I/II Study of Percutaneous Radiofrequency Ablation of Bone Metastases Using CT Guidance
Brief Title: Radiofrequency Ablation in Treating Patients With Bone Metastases
Acronym: ACRIN-6661
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069012; ACRIN-6661 (Other: CIP); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: bone metastases; pain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Analgesia; Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: The outcomes of the study will be adverse event analysis and pain relief.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RFA as pain therapy (Experimental): Changes in the severity of pain as measured using using the Memorial Pain Assessment Cards (MPAC) before and after RadioFrequency Ablation (RFA) will be statistically analyzed
  Interventions: Procedure: pain therapy; Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: pain therapy
Procedure: radiofrequency ablation
  Other Names: RFA

SUMMARY:
RATIONALE: Radiofrequency ablation may be effective in decreasing pain from bone metastases.

PURPOSE: Phase I/II trial to study the effectiveness of radiofrequency ablation in decreasing pain in patients who have bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the side effects of radiofrequency ablation in patients with bone metastases.
* Determine the effect of this regimen on pain in these patients.
* Determine the effect of this regimen on mood in these patients.
* Determine the effects of narcotic usage in patients treated with this regimen.
* Determine the relationship between laboratory and imaging features of this treatment and the effects of the treatment in these patients.

OUTLINE: This is a multicenter study.

Patients undergo percutaneous CT-guided radiofrequency ablation directly to the metastatic lesion over approximately 12 minutes.

Pain and mood are assessed at baseline, daily for 14 days after treatment, and at 1 and 3 months after treatment.

Patients are followed at 1 week and then at 1 and 3 months.

PROJECTED ACCRUAL: Approximately 75 patients will be accrued for this study within 12.5 months.

ELIGIBILITY:
4.1 Inclusion Criteria

4.1.1 Histologically or cytologically documented malignant disease with a bone lesion that has the clinical and/imaging features of metastatic disease.

4.1.2 Persistent intractable pain that results in a return visit to the oncologist. The measurable pain must be above a pain scale of five (scale of 0-10). (Pain during the last week described as "the worst" by the patient on a scale of 0 (no pain) to 10 (pain as bad as patient can imagine)).

4.1.3 The patient's pain must be from a solitary site of metastatic disease in the bone. Each site must be amenable to RFA utilizing a percutaneous CT-guided approach. (RF electrode can be safely placed under CT guidance without harm to normal structures.) 4.1.4 The maximum size of the bone metastasis (study site) must be no greater than 8 cm.

4.1.5 Radiofrequency treatment can be performed within 5 days of baseline evaluations.

4.1.6 All patients must understand and sign a study-specific informed consent.

4.2 Exclusion Criteria

4.2.1 Tumor mass in contact with hollow viscera. 4.2.2 Uncontrolled coagulopathy or bleeding diathesis that cannot be corrected with FFP and platelets prior to procedure. (Platelets must be ≥ 70,000/ul.) 4.2.3 Aspirin and nonsteroidal anti-inflammatory medications, antiplatelet medications, or warfarin must be discontinued prior to the procedure for a time period that is appropriate given the drug half life and the drugs known antiplatelet activity (e.g. aspirin for 7 days and ibuprofen 24 hours). Low molecular weight heparin preparations must be discontinued 24 hours prior to procedure.

4.2.4 Tumor involves a weight-bearing long-bone of the lower extremity. 4.2.5 Site of tumor surgically stabilized with metallic hardware. 4.2.6 Previous (within 30 days immediately prior to RFA or post RFA) or scheduled concurrent systemic treatment of metastases with external beam radiation or radioisotopes. (Chemotherapy will not be allowed within 14 days prior to and within 14 days post RFA procedure).

4.2.7 Patients with primary musculoskeletal malignancies, lymphoma and leukemia will not be RFA treatment candidates.

4.2.8 Spinal metastases that do not have an intact cortex between the mass and the spinal canal and exiting nerve roots.

4.2.8 Patients with a pacemaker.

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2001-11; Primary Completion 2010-02-15 (Actual); Study Completion 2010-02-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | 1 month post procedure
  Estimate the adverse event rate due to RFA within 1 month follow-up period.

SECONDARY OUTCOMES:
Pain intensity | 1 month post-procedure
  pain intensity as measured by VASPI Scale
Pain intensity | 3 months post-procedure
  pain intensity as measured by VASPI Scale
Pain reduction | 1 month post-procedure
  pain reduction as measured by VASPR Scale
Pain reduction | 3 month post-procedure
  pain reduction as measured by VASPR Scale
Mood | 1 month post-procedure
  Mood as measured byt the VASMOOD scale
Mood | 3 month post-procedure
  Mood as measured by the VASMOOD scale
Pain Severity | 1 month post-procedure
  Pain severity as measured by the Tursky scale
Pain Severity | 3 month post-procedure
  Pain severity as measured by the Tursky scale

CONTACTS AND LOCATIONS:
Overall Officials: Damian E. Dupuy, MD, Study Chair — Rhode Island Hospital
Locations (8):
- United States (8):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Mallinckrodt Institute of Radiology at Washington University Medical Center, St Louis, Missouri
  - Radiology Consultants, Incorporated, Youngstown, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Comprehensive Cancer Center at Rhode Island Hospital, Providence, Rhode Island
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All De-identified study data is available to request from ACRIN:
  https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- [Result] Dupuy DE, Liu D, Hartfeil D, Hanna L, Blume JD, Ahrar K, Lopez R, Safran H, DiPetrillo T. Percutaneous radiofrequency ablation of painful osseous metastases: a multicenter American College of Radiology Imaging Network trial. Cancer. 2010 Feb 15;116(4):989-97. doi: 10.1002/cncr.24837. PMID 20041484